CLINICAL TRIAL: NCT05026970
Title: Validation of a Multimodal Algorithm for Treatment of Fecal Incontinence in Women: Study of the Efficacy of the Combination of Treatments on the Impact on Clinical Severity and Quality of Life, and on the Underlying Pathophysiology
Brief Title: Validation of a Multimodal Algorithm for the Treatment of Fecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Lluís Mundet, Motility Unit Coordinator, Hospital de Mataró
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/19
Record Dates: First submitted 2020-04-13; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; anorectal physiology; pragmatic clinical trial
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback+Electrostimulation+Kegel (Active Comparator): Biofeedback (3 sessions) Electrostimulation (12 weeks daily treatment) Kegel exercises (twice daily)
  Interventions: Device: Biofeedback+Tibial Neuromodulation+Kegel; Combination Product: Biofeedback+Kegel
- Biofeedback+Tibial Neuromodulation+Kegel (Active Comparator): Biofeedback (3 sessions) Transcutaneous Neuromodulation (12 weeks daily treatment) Kegel exercises (twice daily)
  Interventions: Combination Product: Biofeedback+Electrostimulation+Kegel; Combination Product: Biofeedback+Kegel
- Biofeedback+Kegel (Active Comparator): Biofeedback (6 sessions) Kegel exercises (twice daily)
  Interventions: Combination Product: Biofeedback+Electrostimulation+Kegel; Device: Biofeedback+Tibial Neuromodulation+Kegel

INTERVENTIONS:
Combination Product: Biofeedback+Electrostimulation+Kegel — Biofeedback (3 sessions) Electrostimulation (12 weeks daily treatment) Kegel exercises (twice daily)
  Other Names: BF+ES+K
  Arms: Biofeedback+Kegel; Biofeedback+Tibial Neuromodulation+Kegel
Device: Biofeedback+Tibial Neuromodulation+Kegel — Biofeedback (3 sessions) Transcutaneous Neuromodulation (12 weeks daily treatment) Kegel exercises (twice daily)
  Other Names: BF+tNM+K
  Arms: Biofeedback+Electrostimulation+Kegel; Biofeedback+Kegel
Combination Product: Biofeedback+Kegel — Biofeedback+Kegel exercises
  Other Names: BF+K
  Arms: Biofeedback+Electrostimulation+Kegel; Biofeedback+Tibial Neuromodulation+Kegel

SUMMARY:
Thisi is a pragmatical clinical trial with the main aim of main aim of evaluating the effectiveness of the combination of treatments for the management of fecal incontinence (FI), on profiles of patients with IF based on pathophysiological criteria, measuring physiological, clinical and quality of life outputs.

Secondary:

1. Evaluate the presence of SIBO, gluten-sensitive enteropathy, malabsorption of bile salts or sugars in patients with Bristol stools ≥5 that condition the fecal continuity.
2. Effect of change in fecal consistency on IF symptoms.
3. To evaluate the effect of the combination of treatments on anorectal physiology and neurophysiology (motor and sensory), clinical severity and quality of life.
4. Evaluate the persistence of the treatments to the three months of end of the same.

DETAILED DESCRIPTION:
FI is a very prevalent condition in community dwelling women. We have previously studied the efectivenes of four treatments in women with FI as well as the effect on the anorectal physiology and neurophysiology. All treatments improved clinical symptoms of FI but there were no statistical differences between the treatments, that were Kegel exercises (K), biofeedback (BF)+K, electrostimulation (ES)+K, and transcutaneous neuromodulation (tNM)+K. With this prevoous study we have a clearer idea of the anorectal physiology which should allow to select patients for given treatments.

For the present study we try to validate a multimodal algorithm to treat FI, taking into account the underlying pahtophysiology.

It will have 2 differentiated stages:

Stage 1: Patients with loose stools (Bristol >5): they will be studied to determine the cause of the diahrrea (mainly food intolerances) and treated accordingly. If FI symptoms remain, patients will pass to:

Stage 2: Patients with Bristol<6 anf FI symptoms. They will be adressed to 3 combinations of treatments according to the pathophysiology that explain the symptoms, which will be:

BF+ES+K: those patients with direct sphincter damage BF+tNM+K: patients with external anal sphincter dennervation and/or colonic motility disorders.

BF alones: patients with FI mainly explained by a bad control of the pelvic floor function (akinesia/dyssynergia).

All patients will be studied with High Resolution Anorectal Manometry, PNTML, endoanal unltrasonography. Clinical severity and QoL with dedicated intruments or questionnaires.

If after 1sr stage, if so, patients have a clinical severity of Cleveland<4 they will be followed up at 3 months with K, studued again their clinical severity and QoL.

After 2nd stage, if so, 3-month of targeted treatment will be performed, and reevaluated with HRAM, PNTML and clinical questionnaires. They will be followed up at 3 monts with only K to study the persistance of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* FI episodes at least 6 months before
* FI episodes each month
* No other treatment the year before
* Able to self-administer treatments

Exclusion Criteria:

* Pregnancy
* If, to investigators criteria, patient will fail to administer the tratmetns properly, due to physical or psychic conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Cleveland Severity Score | 3 month and 6 month
  Changes in clinical severity after the treatments measured with Cleveland score, which ranges from 0 (total continence) to 20 (very severe incontinence)
Anorectal physiology (motor) | 3 month and 6 month
  Changes in anal mean resting pressure and squeeze (voluntary) pressure after the treatments measured with mmHg
Anorectal physiology (sensorial) | 3 month and 6 month
  Changes in rectal sensory thresholds after the treatments measured in volume (milliliters) of rectal distention
Anorectal neurophysiology | 3 month and 6 month
  Changes in pudendal nerve terminal motor latency (PNTML) measured with milliseconds
Quality of Life (QoL) according to FIQL scale | 3 month and 6 month
  Improvements in Fecal incontinence-related QoL after the treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No